CLINICAL TRIAL: NCT03267303
Title: A Phase II, Double-blind, Parallel-group Comparative Study 2 of TS-091 in Patients with Narcolepsy
Brief Title: A Study to Evaluate the Safety and Efficacy of TS-091 in Patients with Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS091-1701; JapicCTI-173689 (Other: JapicCTI)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2019-10

CONDITIONS: Narcolepsy
Keywords: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TS-091 5mg (Experimental)
  Interventions: Drug: TS-091 5mg
- TS-091 10mg (Experimental)
  Interventions: Drug: TS-091 10mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-091 5mg — Orally taken once daily for 3 weeks
  Arms: TS-091 5mg
Drug: TS-091 10mg — Orally taken once daily for 3 weeks
  Arms: TS-091 10mg
Drug: Placebo — Orally taken once daily for 3 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety after administration of TS-091 compared with placebo in patients with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with narcolepsy type 1 or type 2 based on the International Classification of Sleep Disorders, third edition (ICSD-3) criteria
2. Patients aged ≥16 to <65 years at the time of obtaining informed consent
3. Outpatients

Exclusion Criteria:

1. Patients with sleep disorders other than narcolepsy (e.g., sleep apnea syndrome, periodic limb movement disorder)
2. Patients with organic brain diseases (including neurodegenerative diseases or cerebrovascular disorders) or epilepsy
3. Patients with obstructive respiratory diseases (bronchial asthma, emphysema)
4. Patients with psychiatric disorders (e.g., major depressive disorder, bipolar disorder, schizophrenia)

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Mean sleep latency in maintenance of wakefulness test | 3 weeks

SECONDARY OUTCOMES:
Total score on the epworth sleepiness scale | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (2):
- Taisho Pharmaceutical Co., Ltd selected site, Osaka and Other Japanese City, Japan
- Taisho Pharmaceutical Co., Ltd selected site, Seoul and Other Korean City, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inoue Y, Uchiyama M, Umeuchi H, Onishi K, Ogo H, Kitajima I, Matsushita I, Nishino I, Uchimura N. Optimal dose determination of enerisant (TS-091) for patients with narcolepsy: two randomized, double-blind, placebo-controlled trials. BMC Psychiatry. 2022 Feb 22;22(1):141. doi: 10.1186/s12888-022-03785-7. PMID 35193545